CLINICAL TRIAL: NCT01302613
Title: A Pilot and Phase II Study of Altered Chemotherapy Sequencing During Neoadjuvant Therapy for Patients With Stage II or III Rectal Adenocarcinoma
Brief Title: Altered Chemotherapy Sequencing During Neoadjuvant Therapy for Patients With Stage II or III Rectal Adenocarcinoma
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Drug shortage
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU 082010-335
Record Dates: First submitted 2011-02-21; First posted 2011-02-24 (Estimated); Last update posted 2020-08-20 (Actual); Status verified 2019-02

CONDITIONS: Stage II Rectal Cancer; Stage III Rectal Cancer
Keywords: rectal cancer
MeSH Terms: conditions — Rectal Neoplasms | interventions — Capecitabine; Fluorouracil; Leucovorin; Oxaliplatin; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- arm one (Other): RT + Chemo + surgery
  Interventions: Drug: Capecitabine; Drug: 5-FU; Drug: Leucovorin; Drug: Oxaliplatin; Radiation: radiation; Procedure: total mesorectal excision

INTERVENTIONS:
Drug: Capecitabine — Capecitabine will be delivered concurrently with the radiation therapy, at a dose of 1650 mg/m2 divided in even BID doses. It will only be taken on the days of radiation treatment (Monday-Friday, except for holidays). The A.M. dose of the capecitabine must be taken at least one hour prior to the radiation treatment.
Drug: 5-FU — 5-FU 400 mg/m2, iv bolus on day 1 followed by 2400 mg/m2 iv over 46 hours of each cycle. A cycle is delivered every two weeks. Three cycles will be given prior to the surgery. Five additional cycles will be given after surgery.
Drug: Leucovorin — Leucovorin 400 mg/m2, IV, over 2 hours before 5-FU on day 1 of each cycle. A cycle is delivered every two weeks. Three cycles will be given prior to the surgery. Five additional cycles will be given after surgery.
Drug: Oxaliplatin — Oxaliplatin 85mg/m2 IV on day 1 of each cycle. A cycle is delivered every two weeks. Three cycles will be given prior to the surgery. Five additional cycles will be given after surgery.
Radiation: radiation — 28-30 fractions of radiation, given once a day, five days per week (Monday-Friday, except for holidays). The prescribed fraction dose is 180 cGy; the total radiation dose is thus 5040-5400 cGy. The primary treatment fields will be treated with 25 fractions of 180 cGy/fraction with a "boost" of 3-5 fractions of 180 cGy subsequently delivered.
Procedure: total mesorectal excision — Optimal surgical technique involving use of total mesorectal excision (TME) is mandated. The type of surgery, either low anterior resection with sparing of the sphincter mechanism or sphincter-eliminating abdominoperineal resection (APR), will be at the discretion of the attending surgeon.

SUMMARY:
The primary objective of the pilot portion of this study is to establish the safety and tolerability of an extended treatment break period in patients who have undergone neoadjuvant chemoradiotherapy as well as use of systemic therapy during this break.

DETAILED DESCRIPTION:
The proposed protocol aims to continue tumor-directed therapy during the typical "break period" in an effort to improve on both local tumor response as well as distant disease control. First, the duration from completion of chemoradiotherapy would increase from 6-8 weeks to 9-11 weeks. As noted above, this may allow for further cell death with resultant pathologic downstaging. Secondly, the protocol calls for continued systemic therapy during the 9-11 week period, thus allowing continuation of therapies directed towards both the primary as well as distant sites of disease. The primary aim of this pilot study would be to establish the feasibility of this intensified neoadjuvant approach, especially with respect to tolerability of the subsequent pelvic surgery. A subsequent phase II portion will evaluate the efficacy of this treatment approach.

ELIGIBILITY:
Inclusion Criteria:

1. Signed study-specific informed consent form
2. Age > 18 years old
3. Zubrod performance status 0-1
4. Biopsy proven primary malignancy
5. AJCC Stage II or III disease (T3-4 and/or N1-2 disease) as determined by endoscopic ultrasound and/or MRI staging
6. Pretreatment rectal endoscopic ultrasound and pelvic MRI, colonoscopy, CT of chest, abdomen, and pelvis, and laboratory values as discussed below

Exclusion Criteria:

1. History of inflammatory bowel disease
2. Previous pelvic radiotherapy
3. A major psychiatric illness which would limit understanding of the proposed protocol treatment and consent process.
4. Men and women of reproductive potential must agree to use an effective contraception method
5. Pregnant or lactating women
6. Severe, active co-morbidity, defined as

   * Unstable angina and/or CHF requiring hospitalization within the last six months
   * Transmural myocardial infarction within the last 6 months
   * Acute bacterial or fungal infection requiring intravenous antibiotics at the time of registration
7. Presence of metastatic disease, including liver metastases
8. Laboratory values out of range

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-03; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
The primary study endpoint for the phase I portion of this study is to assess surgical complications through the Clavien grading system. | 90 days
  The adverse events will be followed prospectively from the date of surgery for 90 days. Dose-limiting toxicity (DLT) will be defined as > grade 3 anastomotic stricture or leak, infection (including pelvic abscess or wound infection), small bowel obstruction, or fistualization. Any other post-operative complication thought related directly to the surgical intervention that is a grade 3 or higher Clavien complication will also be considered dose-limiting toxicity.

SECONDARY OUTCOMES:
The primary endpoint of the phase II portion of the study is complete pathologic response. | 9 to 11 weeks
  9 to 11 weeks after the completion of the initial chemoradiotherapy.

CONTACTS AND LOCATIONS:
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States